CLINICAL TRIAL: NCT02543073
Title: Mesenchymal Stem Cell for Treatment of Interstitial Lung Disease After Allogenetic Hematopoietic Stem Cell Transplantation
Brief Title: MSC for Treatment of Interstitial Lung Disease After Allo-HSCT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-ILD-2015
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2015-09

CONDITIONS: Lung Diseases, Interstitial; Hematopoietic Stem Cell Transplantation; Bronchiolitis Obliterans
MeSH Terms: conditions — Lung Diseases, Interstitial; Bronchiolitis Obliterans | interventions — Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSCs (Experimental): MSCs will be given the patients in MSCs group. Besides, azithromycin (AZM) and glucocorticoid will also be administered.
  Interventions: Biological: MSCs; Drug: AZM; Drug: Glucocorticoid
- Non-MSCs (Active Comparator): AZM and glucocorticoid will be given for the patients in Non-MSCs group.
  Interventions: Drug: AZM; Drug: Glucocorticoid

INTERVENTIONS:
Biological: MSCs — MSCs will be given at a median dose of 1×10^6 cells/kg once weekly for 4 weeks as one cycle treatment.
  Arms: MSCs
Drug: AZM — AZM will be given （0.25g qd）for 4 weeks as one cycle treatment.
Drug: Glucocorticoid — Glucocorticoid (prednison) will be given at the starting dose of 1mg/kg for 4 weeks as one cycle treatment.

SUMMARY:
Interstitial lung disease (ILD） is the late pulmonary complications after allogeneic hematopoietic stem cell transplantation (allo-HSCT) leading to high morbidity and mortality. At present, the treatment for ILD after allo-HSCT remains in discussion. In this study, the efficacy of mesenchymal stem cells (MSCs) combined azithromycin as well as glucocorticoid as the treatment of ILD will be evaluated in the recipients of allo-HSCT.

DETAILED DESCRIPTION:
ILD is a group of diseases involving pulmonary interstitial, alveolar and (or) bronchioles. In the patients receiving allo-HSCT, ILD mainly present as bronchiolitis obliterans syndrome (BOS). ILD after HSCT is characterized by non-responsiveness to treatment, leading to high morbidity and mortality. MSC has been considered as an effective treatment for refractory acute graft-versus-host disease (aGVHD), but the response to treat chronic GVHD (cGVHD), especially refractory BOS, is rarely reported.

ELIGIBILITY:
Inclusion Criteria:

* Receiving allo-HSCT
* Diagnosed with ILD after allo-HSCT

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Response rate of ILD | 4 weeks
  Response includes complete response (CR) and partial response (PR). CR is defined as resolution of all manifestations related to ILD, except for some irreversible changes. PR is defined as sustained, measurable improvement in pulmonary function tests(carbon monoxide lung diffusion capacity, forced expiratory volume, or both) or the ability to reduce corticosteroids by at least 50% or both without deterioration of pulmonary function.

SECONDARY OUTCOMES:
Overall Survival | 3 year
  The 3-year overall survival after HSCT will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Olivieri A, Locatelli F, Zecca M, Sanna A, Cimminiello M, Raimondi R, Gini G, Mordini N, Balduzzi A, Leoni P, Gabrielli A, Bacigalupo A. Imatinib for refractory chronic graft-versus-host disease with fibrotic features. Blood. 2009 Jul 16;114(3):709-18. doi: 10.1182/blood-2009-02-204156. Epub 2009 Apr 29. PMID 19403889
- [Derived] Chen S, Zhao K, Lin R, Wang S, Fan Z, Huang F, Chen X, Nie D, Du X, Guo Z, Lin D, Xuan L, Xu N, Sun J, Peng Xiang A, Liu Q. The efficacy of mesenchymal stem cells in bronchiolitis obliterans syndrome after allogeneic HSCT: A multicenter prospective cohort study. EBioMedicine. 2019 Nov;49:213-222. doi: 10.1016/j.ebiom.2019.09.039. Epub 2019 Oct 23. PMID 31668569